CLINICAL TRIAL: NCT07251296
Title: Effects of a Nutritional Supplement and Physical Exercise on the Psycho-emotional, Cognitive, Functional, and Neuroendocrine Health of Perimenopausal Women.
Brief Title: Impact of Funcional Exercise and Supplementation in Perimenopausal Women's Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan C. Colado, Professor of Physical Education, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-FIS-4025659
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Perimenopause; Aging
Keywords: Perimenopause; nutritional supplement; Functional exercise; Psycho-emotional health; Cognitive function; Non-pharmacological interevention; Randomized controlled trial; Physical function; variable resistance training; Neuroendocrine biomarkers; Sleep and mood regulation
MeSH Terms: interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + nutritional supplement (Gr 1: EXNS) (Experimental): Participants in this group will receive a daily dose of the natural-origin nutritional supplement in combination with a supervised functional exercise program (3 sessions per week, 45-60 minutes each) for 10 weeks.
  Interventions: Dietary Supplement: Exercise + nutritional supplement
- Exercise + placebo supplement (Gr 2: EXPLA) (Placebo Comparator): Participants in this group will receive a placebo supplement identical in appearance to the active supplement, together with the same functional exercise program for 10 weeks.
  Interventions: Dietary Supplement: Exercise + placebo supplement

INTERVENTIONS:
Dietary Supplement: Exercise + nutritional supplement — Participants in this group will receive an oral daily dose of the natural-origin nutritional supplement in combination with a supervised functional exercise program (3 sessions per week, 45-60 minutes each) for 10 weeks, composed by three exercise blocks: 1) joint mobility and postural control exercises block, 2) functional strength block with three sets of two explosive strength exercises using elastic bands at 70% of 1RM and, 3) coordination and agility exercises block.
  Arms: Exercise + nutritional supplement (Gr 1: EXNS)
Dietary Supplement: Exercise + placebo supplement — Participants in this group will receive an oral placebo supplement identical in appearance to the active supplement, together with the same functional exercise program for 10 weeks.
  Arms: Exercise + placebo supplement (Gr 2: EXPLA)

SUMMARY:
The goal of this clinical trial is to learn whether a natural-origin nutritional supplement, combined with a functional exercise program, can improve psycho-emotional, cognitive, functional, and neuroendocrine health in perimenopausal women. The study will also help determine the safety of this combined intervention.

The main questions it aims to answer are:

* Does the combined intervention improve mood, sleep quality, menopausal symptoms, and cognitive performance?
* Does it enhance physical function and neuroendocrine regulation?

Researchers will compare the supplement to a placebo. All participants will follow the same supervised functional exercise program.

Participants will:

* Take a daily nutritional supplement or placebo for 10 weeks
* Attend three weekly supervised functional exercise sessions (45-60 minutes each)
* Complete pre- and post-intervention evaluations including questionnaires, physical and cognitive tests, and blood samples for biomarker analysis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial with parallel groups, designed to evaluate the effects of a natural-origin nutritional supplement combined with a functional physical exercise program on psycho-emotional, cognitive, functional, and neuroendocrine variables in perimenopausal women. Participants will be randomly assigned to the intervention groups, with both participants and outcome assessors blinded to group allocation (double-blind design). All study groups will receive a functional exercise intervention, in addition to the nutritional supplement or placebo.

The study will last a total of 10 weeks and will include a supervised functional exercise program consisting of three weekly sessions, each lasting 45 to 60 minutes. Pre- and post-intervention assessments will be conducted, including validated questionnaires on sleep quality, mood, general well-being, and menopausal symptoms; objective cognitive tests (attention, working memory, and executive functions); physical fitness assessments (strength, agility, gait speed, body composition); and blood analyses of neuroendocrine biomarkers (cortisol, BDNF, IL-6, TNF-α, GABA, and serotonin).

This methodological design will allow for both within- and between-group comparisons and the analysis of potential interactions between the interventions, in order to determine their efficacy and safety as non-pharmacological strategies to improve the overall health of perimenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 45 and 65 years.
* In the menopausal transition (defined by irregular menstrual cycles and typical symptoms within the past year) or postmenopause.
* Score ≥ 8 on the Menopause Rating Scale (MRS), indicating moderate menopausal symptom intensity.
* Regular nighttime sleep and not engaged in shift work.
* Low physical activity level: less than 150 minutes per week of moderate or vigorous physical activity, as assessed by the short-form IPAQ or a similar questionnaire.
* Body mass index (BMI) between 18.5 and 35 kg/m².
* Sufficient functional and cognitive capacity to participate in supervised physical exercise and follow the study protocol.
* Signed informed consent and availability to attend all scheduled sessions and assessments.

Exclusion Criteria:

* Current or recent (within the last 3 months) use of hormone replacement therapy (HRT).
* Surgical, induced, or early menopause (before age 40).
* Current treatment with medications that may affect mood, sleep, or vasomotor symptoms, including: antidepressants (SSRIs, SNRIs, tricyclics); anxiolytics or hypnotics; phytoestrogens, isoflavones, or other over-the-counter hormonal supplements.
* Medical diagnosis of severe or uncontrolled chronic diseases, including cardiovascular, respiratory (particularly sleep apnea), metabolic, active oncological, neurological, severe autoimmune, or psychiatric disorders.
* Regular use within the past 3 months of nutritional or sports supplements that may interfere with study outcomes (e.g., creatine, protein, omega-3, adaptogens, etc.).
* Medical contraindications for moderate-to-vigorous physical exercise, as determined by the PAR-Q+ questionnaire and/or updated medical report.
* Simultaneous participation in another clinical trial or intervention program involving drugs, supplements, or structured physical exercise of any kind.
* Known allergy or intolerance to any component of the nutritional supplement to be administered.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Brain-Derived Neurotrophic Factor (BDNF) | Before and after the intervention of 10 weeks
  Serum BDNF levels will be collected through a blood sample (ELISA KIT) in the morning in a fasted state to assess neuroplasticity and cognition.
Changes in cortisol | Before and after the intervention of 10 weeks
  Serum cortisol levels will be collected through a blood sample (ELISA KIT) in the morning in a fasted state to assess hypothalamic-pituitary-adrenal (HPA) axis-mediated physiological stress.
Changes in inteleukin 6 (IL-6) | Before and after the intervention of 10 weeks
  Serum IL-6 levels will be collected through a blood sample (ELISA KIT) in the morning in a fasted state to assess systemic inflammation and immunity
Changes in tumor necrosis factor alfa (TNF-α) | Before and after the intervention of 10 weeks
  Serum TNF-α levels will be collected through a blood sample (ELISA KIT) in the morning in a fasted state to assess chronic inflammation and immune state, which is related with fatigue and depression.
Changes in Gamma-aminobutyric acid (GABA) | Before and after the intervention of 10 weeks
  Serum GABA levels will be collected through a blood sample (ELISA KIT) in the morning in a fasted state to assess the state of the central nervous system, related with relaxation, anxiety and sleep conditions.
Changes in serotonin | Before and after the intervention of 10 weeks
  Serum serotonin levels will be collected through a blood sample (ELISA KIT) in the morning in a fasted state as a key neurotransmitter involved in mood regulation, sleep, and cognition.

SECONDARY OUTCOMES:
Changes in sleep quality | Before and after the intervention of 10 weeks
  Sleep quality will be assessed through the Pittsburgh Sleep Quality Index (PSQI)
Changes in perceived insomnia | Before and after the intervention of 10 weeks
  Perceived insomnia will be assessed through the Insomnia Severity Index (ISI)
Changes in daytime sleepiness | Before and after the intervention of 10 weeks
  Daytime sleepiness will be assessed through the Epworth Sleepiness Scale (ESS)
Changes in state-trait anxiety | Before and after the intervention of 10 weeks
  State-trait anxiety will be assessed through the State-Trait Anxiety Inventory (STAI-R)
Change in depression | Before and after the intervention of 10 weeks
  Depression will be assessed through the Beck Depression Inventory-II (BDI-II)
Changes in general well-being | Before and after the intervention of 10 weeks
  General well-being will be assessed through the WHO-5 Well-Being Index
Changes in menopausal symptoms | Before and after the intervention of 10 weeks
  Menopausal symptoms will be assessed through the Menopause Rating Scale (MRS)
Changes in global cognitive performance | Before and after the intervention of 10 weeks
  Global cognitive performance will be assessed through the Montreal Cognitive Assessment (MoCA)
Changes in working memory | Before and after the intervention of 10 weeks
  Working memory will be assessed through the Digit Span (WAIS-IV Digit Span subtest - forward and backward)
Changes in selective attention | Before and after the intervention of 10 weeks
  Selective attention will be assessed through the Stroop Test (short version)
Changes in processing speed and cognitive flexibility | Before and after the intervention of 10 weeks
  Processing speed and cognitive flexibility will be assessed through the Trail Making Test A and B (TMT-A/B)
Changes in gait speed/aerobic capacity | Before and after the intervention of 10 weeks
  Gait speed/aerobic capacity will be assessed through the 6-m Walk Test
Changes in lower limb strength | Before and after the intervention of 10 weeks
  Lower limb strength will be assessed through the 30-s Chair Stand Test
Changes in handgrip strength | Before and after the intervention of 10 weeks
  Handgrip strength will be assessed through the Handgrip dynamometry (Jamar Hand Dynamometer).
Changes in body composition | Before and after the intervention of 10 weeks
  Whole body composition will be assessed through the Bioelectrical impedance analysis (Tanita BC-418). Total body mass, fat mass, fat-free mass and percentage of fat free mass will be measured.
Adherence to supplement and exercise | Every day for nutritional supplement and each exercise session during the 10 weeks of intervention
  Adherence to supplement and exercise will be assessed through ad hoc questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Physical activity and Sport Science Faculty, Valencia, Valencia 46010, Valencia, Valencia, Spain